CLINICAL TRIAL: NCT04728997
Title: Reliability and Validity of the Turkish Version of the Abiloco
Brief Title: Mobility Assessment in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Keski̇n, Research Asistant, MSc, Hacettepe University
Other Study IDs: EKeskin
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Stroke
Keywords: stroke, questionnaire, ABILOCO
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Stroke ranks 3rd among disability-causing diseases worldwide. Following a stroke, loss of lower extremity motor function causes serious gait disturbances. The walking activity is the basis for daily and social engagement activities. Mobility (locomotion) ability; gait analysis can be evaluated with tests and reports examining walking performance. ABILOCO is also a questionnaire developed by Caty et al., evaluating mobility and locomotion in individuals after stroke. The aim of this study is; To investigate the validity and reliability of the Turkish version of the ABILOCO questionnaire developed to evaluate mobility in patients with stroke. The sample of the study will be literate individuals who have had a stroke who applied to the Neurology Unit of Ankara Hacettepe University Faculty of Physical Medicine and Rehabilitation.

Demographic information of the cases will be recorded. ABILOCO questionnaire will be adapted to Turkish. The validity and reliability comparison of the ABILOCO questionnaire with the Berg Balance Scale and Timed Get Up and Go Test will be performed.

DETAILED DESCRIPTION:
The sample of the study will consist of literate individuals who applied to Ankara Hacettepe University Faculty of Physical Medicine and Rehabilitation, Physiotherapy and Rehabilitation Department and were diagnosed with stroke. The number of cases in the study will be determined as 5 to 10 times the number of items in the questionnaire, and 65-130 individuals will be included.

Inclusion Criteria:

* Having a definite stroke diagnosis
* Those who have stable post-stroke systemic findings
* Mini-mental test score of 24 and above
* Those who can walk 10 meters unsupported
* Those who passed 2 months after stroke.

Criteria for exclusion from the study:

- Having musculoskeletal problems that affect the mobility of the individual.

The study will use ABILOCO, which has been validated for individuals with stroke. Permission was obtained from Gilles D. Caty, the development of the questionnaire, to conduct translation and validity and cultural adaptation stduies into Turkish. In the study, firstly, the original English version of the questionnaire will be translated into Turkish by two professional translators independent of the study, and then it will be translated back into its original language English by two native English speakers who do not have a medical background. Translators will be brought together to discuss the two obtained versions of the questionnaire. The latest version of the questionnaire will be translated into the native language of the inventory and its compliance will be checked. Mini-Mental Test will be applied to determine the cognitive status of the participants. Berg Balance Scale and Timed Get Up and Go Test will be applied for mobility assessment. After that, the ABILOCO questionnaire will be applied to the participants. In order to test the reliability of the survey, the survey will be repeated 7 days later. Informed consent will be obtained from each participant regarding their voluntary participation in the study and their sociodemographic information will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* having a definite stroke and have passed 2 months post-stroke
* individuals who can walk 10 meters without support
* Those whose systemic findings are stable after stroke
* Mini-mental test score of 24 and above

Exclusion Criteria:

* Those with musculoskeletal system problems that will affect the individual in terms of mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample of the study will be composed of literate individuals who applied to Ankara Hacettepe University Faculty of Physical Therapy and Rehabilitation, Physiotherapy and Rehabilitation Department and were diagnosed with stroke. The number of cases in the study will be determined as 5 to 10 times the number of items in the questionnaire, and 65-130 individuals will be included.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
ABILOCO Questionnaire | baseline
  Turkish version of ABILOCO questionnaire evaluation of validity and reliability in stroke patients ABILOCO: A questionnaire evaluating mobility

SECONDARY OUTCOMES:
Berg Balance Scale | baseline
  Berg Balance Scale: An assessment evaluating balance and risk of falling
Time up and Go test | baseline
  Time up and Go: A test evaluating mobility (locomotion), requires static and dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: ESRA KESKİN, Principal Investigator — Study Principal İnvestigator
Locations (1):
- Hacettepe Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided